CLINICAL TRIAL: NCT01418742
Title: SKIP - A Double-blind Placebo-controlled Randomized Multicenter Phase II Trial of Skin Toxicity Treatment in Subjects With Advanced or Metastatic Colorectal Carcinoma Receiving Panitumumab
Brief Title: SKIP - A Double-blind Placebo-controlled Randomized Multicenter Trial of Skin Toxicity Treatment
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitement did not meet expectations. Prev. differentiation of RAS-wild-type and mutated RAS are not in accordance with the scientific rank anymore.
Sponsor: Gesellschaft fur Medizinische Innovation - Hamatologie und Onkologie mbH (Other)
Collaborators: ClinAssess GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GMIHO-010/2009
Record Dates: First submitted 2011-08-03; First posted 2011-08-17 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2013-03

CONDITIONS: Colorectal Carcinoma
Keywords: skin toxicity
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Panitumumab; Doxycycline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Doxycycline 100 mg BID oral use (Active Comparator)
  Interventions: Drug: Panitumumab, Doxycycline/Placebo
- Placebo 100 mg BID oral use (Placebo Comparator)
  Interventions: Drug: Panitumumab

INTERVENTIONS:
Drug: Panitumumab, Doxycycline/Placebo — comparison of Doxycyline/Placebo and Panitumumab regarding efficacy of the therapy of panitumumab induced skin toxicity
  Arms: Doxycycline 100 mg BID oral use
Drug: Panitumumab — mCRC patients receiving panitumumab as EGFR inhibitor.
  Arms: Placebo 100 mg BID oral use

SUMMARY:
Skin toxicity treatment in patients with advanced or metastatic colorectal cancer (mCRC) and non-mutated (wild-type) KRAS treated with panitumumab monotherapy after failure of fluoropyrimidine-, oxaliplatin-, and irinotecan-containing chemotherapy regimens.

DETAILED DESCRIPTION:
Because of their frequency and severity panitumumab associated skin toxicities affect patients' quality of life and thus threaten patients' compliance to therapy. There is an urgent need for evidence-based treatment recommendations for the prevention and management of panitumumab -associated skin toxicities.

The study aims to compare the efficacy and safety of a manageable preemptive treatment with oral doxycycline in combination with a supportive topical regimen containing erythromycin cream (2 %) over duration of 12 weeks on the occurrence and grade of panitumumab induced skin toxicities in a double-blind, controlled randomized setting. Basic skin treatment with or without doxycycline will be discontinued at the end of study treatment after 12 weeks or until a value of 6-10 is observed on the visual analogue scale (VAS), whichever is sooner.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced or metastatic colorectal cancer (mCRC) and non-mutated (wild-type) KRAS who are planned to receive treatment with panitumumab monotherapy after failure of fluoropyrimidine-, oxaliplatin-, and irinotecan-containing chemotherapy regimens and without prior treatment with epidermal growth factor receptor (EGFR) antibody
2. Man or woman 18 years of age or older
3. Signed and dated informed consent before the start of specific protocol procedures
4. ECOG (Eastern Cooperative Oncology Group) performance status of 0, 1, or 2
5. Bilirubin ≤ 1.5 x ULN, SGOT/SGPT ≤ 2.5 x ULN, AP ≤ 3 x ULN if no evidence of liver metastases or Bilirubin ≤ 3 x ULN, SGOT/SGPT ≤ 5 x ULN, AP ≤ 5 x ULN if evidence of liver metastases
6. Women of child-bearing potential have to use adequate highly effective methods of contraception . Since doxycyline may reduce efficacy of hormonal contraceptives, women of child-bearing potential have to use double-barrier methods within 4 weeks before first intake of study medication, during study participation and at least 6 weeks after last intake of study medication even if using hormonal contraceptives Women are considered to be of child-bearing potential unless they are ≥ 50 years old and for more than 2 years amenorrheic or unless they are surgically sterile.

Exclusion Criteria:

1. Absence of any of the above-listed inclusion criteria
2. Any serious medical condition or psychiatric illness that would interfere with the patient's ability to sign the informed consent form.
3. Allergic reaction to one of the medications to be used
4. Subject allergic to panitumumab or any components of the panitumumab formulation or treatment regimen
5. Prior treatment with EGFR antibody
6. CYP3A4 enzyme inducers, inhibitors, and substrates (eg, phenytoin, phenobarbital, carbamazepine, ketoconazole, rifampicin, rifabutin, and St. John's Wort) ≤ 2 weeks before randomization (itraconazole should be used with caution)
7. Subjects with hypersensitivity to doxycycline, other tetracyclines, or ingredients of doxycycline capsules
8. Systemic treatment with antibiotics which was completed less than 7 days prior to randomization
9. Pregnant and/or breast-feeding women
10. Active participation in other clinical studies in the previous 4 weeks
11. Serious liver function disorders
12. History of, or evidence of, interstitial pneumonitis or pulmonary fibrosis
13. Person who has been committed to an institution by virtue of an order issued either by the judicial or the administrative authorities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Time until unblinding of skin therapy allocation (basic skin treatment with or without doxycycline) due to insufficient efficacy (i.e. unbearable skin toxicity, measured by patient's allocating point 6 through 10 on a visual analogue scale) | 30 month

SECONDARY OUTCOMES:
Incidence of specific ≥ grade 2 skin toxicities over 12 weeks or until a value of 6-10 is observed on the VAS, whichever is sooner | 30 months
Time to first occurrence of specific ≥ grade 2 skin toxicities | 30 months
Most severe specific ≥ grade 3 skin toxicities of interest over 12 weeks or until a value of 6-10 is observed on the VAS, whichever is sooner | 30 months
Time to the first most severe specific ≥ grade 3 skin toxicities | 30 month
Incidence of panitumumab dose reduction due to the specific skin toxicities of interest over 12 weeks or until a value of 6-10 is observed on the VAS, whichever is sooner | 30 month
Scores in DLQI under preemptive basic skin treatment with or without doxycycline | 30month
Incidence of doxycycline related adverse events | 30 month
Type of panitumumab related adverse events | 30 month
Response rate to panitumumab over 12 weeks or until a value of 6-10 is observed on the VAS, whichever is sooner (only if patient received at least 8 weeks of study treatment) | 30 month
Type of doxycycline related adverse events | 30 month
Severity of doxycycline related adverse events | 30 month
Incidence of panitumumab related adverse events | 30 month
Severity of panitumumab related adverse events | 30 month

CONTACTS AND LOCATIONS:
Overall Officials: Hanno Riess, Prof., Study Chair — Charité Campus Virchow Klinikum, Klinik für Innere Medizin mit Schwerpunkt Hämatologie u. Onkologie
Locations (12):
- Germany (12):
  - DRK Kliniken Berlin / Köpenick, Klinik für Chirurgie, Berlin
  - Onkologische Schwerpunktpraxis, Berlin
  - Medizinisches Versorgungszentrum Ärzteforum Seestraße, Berlin
  - Charité Campus Virchow Klinikum (CVK), Centrum für Tumormedizin, Medizinische Klinik mit Schwerpunkt Hämatologie u. Onkologie, Berlin
  - Ärzteforum Bernau, Bernau
  - Onkologische Schwerpunktpraxis, Brandenburg
  - Städtisches Klinikum Dessau, Hömatologie und Internistische Onkologie, Dessau
  - St. Georg Klinikum Eisenach gGmbH, Klinik für Innere Medizin 2, Eisenach
  - Krankenhaus St. Elisabeth u. St. Barbara, Klinik für Allgemein- u. Visceralchirurgie, Halle
  - Ärzteforum Hennigsdorf, Hennigsdorf
  - eps-early phase GmbH, Jena
  - Klinikum Dorothea Christiane Erxleben Quedlinburg gGmbH, Klinik f. Allgemein, Vizeral- und Gefäßchirurgie, Quedlinburg